CLINICAL TRIAL: NCT01467102
Title: euCPSP: European Observational Study on Chronic Post Surgical Pain,PAIN-OUT
Brief Title: euCPSP: European Observational Study on Chronic Post Surgical Pain,PAIN-OUT Study
Acronym: PAIN-OUT
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Collaborators: University of Jena (Other)
Responsible Party: Sponsor
Other Study IDs: euCPSP PAIN-OUT
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Postoperative Pain
Keywords: chronic post surgical pain; Pain; Risk factors of chronic post surgical pain; predictive risk factors; chronic post-surgical pain (CPSP); international level; epidemiology of CPSP; Europe; observational; prospective
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: > 18 years of age

SUMMARY:
This project a European observational study on the incidence and characteristics of chronic post surgical pain (CPSP).

Research Questions

* What is the incidence of chronic post surgical pain (CPSP) in Europe?
* What are the risk factors of chronic post surgical pain (CPSP) related to surgery, patient and anaesthesia management?
* What are the difference in incidence and risk factors in different European countries?

DETAILED DESCRIPTION:
The main goal of the study is to obtain a generalizable epidemiology of chronic post surgical pain (CPSP) by performing a large data collection in many European countries. The large sample will allow analysis of the incidence of CPSP, differences in incidence patterns in Europe, incidence in rare types of surgeries and specific populations. This observational, prospective study will help to better anticipate and potentially prevent the development of chronic post surgical pain (CPSP). In fact when CPSP occurs patients are frequently undiagnosed and pain is poorly managed such that patients may develop refractory chronic pain. Surgery is a major cause of chronic pain and it is unique in that there is potential to prevent it from occurring. Data from this study might alert respectively surgeons and anesthetists about the most important types of surgery and some perioperative techniques of pain prevention with an impact on the incidence of chronic post surgical pain(CPSP). Anesthesiologists, who are leading this project, might therefore, have an important role in preventing future cases of chronic post surgical pain (CPSP).

Sample size calculation:

The investigators expect that at least 30 sites will be able to participate and recruit 200 patients a year, to a maximum of 6,000 patients, over the one year study period. Since the mean incidence of CPSP is approximately 30%, this will offer an estimated potential number of 2000 patients with CPSP.

Organisation:

Investigators will use questionnaire in English, German, French, Spanish, Italian, Romanian, Swedish, Hebrew, Dutch and Russian. They will supervise data collection, ensure timely data return and act as guarantor for the integrity and quality of data collected.

The Chief investigator, Professor Fletcher is a member of the PAIN OUT group and will closely work with the new group of investigators participating in the project on CPSP. His experience with the European PAIN OUT project will be very valuable to organize and coordinate the study. The European Society of Anaesthesiology (ESA) is supporting this project and will help with administrative coordination to build the European network.

Time scale:

The study will last two and a half years with one year for recruitment, one year for follow up and 6 months for analysis.

Statistical Analysis:

Incidence of chronic post surgical pain (CPSP) at 12 months for all types of surgeries analyzed will be expressed as mean and confidence interval 95%. The investigators will compare the incidence in various types of surgeries, different centres and countries.

Risk factors of chronic post surgical pain (CPSP) will be analyzed using univariate and multivariate analysis. The most predictive factors will be chosen by fitting a logistic regression model using a forward selection procedure. By combining data from different centres, the investigators will determine most significant risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years old and above
* Patient has given consent
* Patient is able to fill in questionnaire on his\her own, unaided (exceptions are patients who are unable to fill in the questionnaire for technical reasons, e.g. can not write due to the surgery (e.g. their arm in a cast) or unable to see the text (e.g. spectacles not available); patient is in department, available for interview.
* Patient is capable of participating in the CPSP incidence study (i.e. capable to fill the questionnaires on the website at 6 and 12 months after surgery).
* Time of data collection immediately after surgery is POD1 and 24±12 hrs after surgery.
* Patient has not undergone repeat surgery (same organ) during current hospitalization.
* Patient has undergone a surgery included in the appendix 1 list below:

List of surgeries to be included:

Surgery without preoperative pain

1. Thoracotomy for lung cancer
2. Breast surgery for cancer
3. Inguinal hernia repair (laparoscopic)
4. Hysterectomy (laparoscopic)
5. Hysterectomy (open)
6. Hysterectomy (vaginal)
7. Colectomy (laparoscopic)
8. Colectomy (open)
9. Thyroidectomy
10. C section
11. High gastric bypass
12. Laparoscopy
13. Prostatectomy

Surgery with potential preoperative pain

1. Cholecystectomy (laparoscopic)
2. Cholecystectomy (open)
3. Total knee arthroplasty
4. Knee arthroscopy
5. Total hip arthroplasty
6. Extracorporeal circulation auxiliary to open heart surgery
7. Spinal surgery
8. Hip arthrotomy

Exclusion Criteria:

* patient not fulfilling at least one of the inclusion criteria mentioned above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient 18 years old and above Patient from European centres Patient able to fill in questionnaire on his\her own, unaided (for exception see protocol) Patient is capable of participating in the CPSP incidence study (i.e. capable to fill the questionnaires on the website at 6 and 12 months after surgery).
  Patient has not undergone repeat surgery (same organ) during current hospitalization.
  Patient has undergone a surgery included in the list of surgeries(see list in eligibility criteria)
Sampling Method: Non-Probability Sample
Enrollment: 3618 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The incidence of chronic post surgical pain (CPSP)12 months after surgery | 12 months
  All patients will be asked to fill the Brief Pain Inventory (BPI) and questionnaires, at 12 months after surgery. They will do it directly on a dedicated website.

SECONDARY OUTCOMES:
Incidence of chronic post surgical pain (CPSP) 6 months after surgery | 6 months
  All patients will be asked to fill the Brief Pain Inventory (BPI) and questionnaires, at 6 months after surgery. They will do it directly on a dedicated website.
risk factors of chronic post surgical pain (CPSP) related to the patient, surgery, anaesthesia and analgesia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Esther Pogatzki-Zahn, MD, Principal Investigator — University Hospital Münster UKM, Munster; Ruth Zaslansky, MD, Principal Investigator — Friedrich Schiller University Jena, Germany; Winfried Meissner, MD, Principal Investigator — Friedrich Schiller University Jena, Germany; Dominique Fletcher, MD, Study Chair — Hôpital Raymond Poincaré AP-HP,Université Versailles St Quentin,Garches, France
Locations (24):
- Belgium (2):
  - Clinique Universitaire de St Luc, Brussels
  - UZA, University Hospital Of Antwerp, Edegem
- Hopital Raymond Poincare, Garches, France
- Germany (3):
  - University Hospital Jena, Jena
  - University Hospital Münster UKM, Münster
  - University of Wuerzburg, Würzburg
- Cork University Hospital, Cork, Ireland
- Italy (2):
  - Policlinico "Oo. Riuniti", Foggia
  - Ii Universita Di Napoli (Policlinico), Napoli
- National Centre of Emergency Medicine, Chisinau, Moldova
- Romania (2):
  - Emergency Institute of Cardiovascular Diseases Inst. '' Prof. C. C . Iliescu'', Bucharest
  - Central Universitty and Emergency Military Hospital "Dr. Carol Davila", Bucharest
- Spain (2):
  - Hospital Universitario de San Juan, Alicante
  - Hospital Del Mar, Barcelona
- Switzerland (5):
  - Inselspital Universitätsklinikum, Bern
  - Hôpitaux Universitaires de Genève, Geneva
  - Lausanne University Hospital, Lausanne
  - Ensemble Hospitalier de la Cote in Morges, Morges
  - Stadtspital Triemli, Zurich
- Ukraine (3):
  - National Cancer Institute, Kiev
  - City Clinical Hospital, Kyiv
  - Zhitomir Regional Oncological centre, Zhytomyr
- United Kingdom (2):
  - Torbay Hospital, Torquay, Devon
  - University College Hospital NHS Foundation Trust, London

REFERENCES:
- [Background] Fletcher D, Pogatzki-Zahn E, Zaslansky R, Meissner W; Pain Out Group. euCPSP: European observational study on chronic post-surgical pain. Eur J Anaesthesiol. 2011 Jun;28(6):461-2. doi: 10.1097/EJA.0b013e328344b4cd. No abstract available. PMID 21544026
- [Derived] Fletcher D, Stamer UM, Pogatzki-Zahn E, Zaslansky R, Tanase NV, Perruchoud C, Kranke P, Komann M, Lehman T, Meissner W; euCPSP group for the Clinical Trial Network group of the European Society of Anaesthesiology. Chronic postsurgical pain in Europe: An observational study. Eur J Anaesthesiol. 2015 Oct;32(10):725-34. doi: 10.1097/EJA.0000000000000319. PMID 26241763
- [Derived] Stamer UM, Naef N, Porz R, Stuber F, Leva B, Meissner W, Fletcher D; euCPSP Study Group. Ethical procedures and patient consent differ in Europe. Eur J Anaesthesiol. 2015 Feb;32(2):126-31. doi: 10.1097/EJA.0000000000000206. PMID 25503525
- See also: PAIN OUT INTERNATIONAL website — http://www.pain-out.eu/